CLINICAL TRIAL: NCT03942601
Title: Temsirolimus Alone or Paired With Dexamethasone Delivered to the Adventitia to eNhance Clinical Efficacy After Femoropopliteal Revascularization
Acronym: TAP-DANCE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Halted due to pandemic.
Sponsor: Mercator MedSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIP0215
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — temsirolimus; dexamethasone 21-phosphate

STUDY DESIGN:
Intervention Model Description: This is an open-label study without randomization. Cohorts will be enrolled sequentially, with Group 1 followed by Group 2.
  Study Drug: Temsirolimus Injection (0.4 mg/mL) and 20% contrast in Group 1 or Temsirolimus Injection (0.4 mg/mL), Dexamethasone Sodium Phosphate Injection, USP (3.2 mg/mL) and 20% contrast in Group 2 Route of Administration: Bullfrog Micro-Infusion Device adventitial delivery Dosage Volume:0.5 mL per cm of target vessel length Up to 30 subjects in Group 1 and up to 30 subjects in Group 2. The study shall enroll subjects from up to 20 sites in the United States.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 - temsirolimus injection (Active Comparator): Temsirolimus Injection (0.4 mg/mL) and 20% contrast in Group 1
  Interventions: Drug: Temsirolimus
- Group 2 - temsirolimus and dexamethasone injection (Active Comparator): Temsirolimus Injection (0.4 mg/mL), Dexamethasone Sodium Phosphate Injection, USP (3.2 mg/mL) and 20% contrast in Group 2
  Interventions: Drug: Temsirolimus and dexamethasone sodium phosphate

INTERVENTIONS:
Drug: Temsirolimus — Temsirolimus Injection (0.4 mg/mL) and 20% contrast in Group 1
  Arms: Group 1 - temsirolimus injection
Drug: Temsirolimus and dexamethasone sodium phosphate — Temsirolimus Injection (0.4 mg/mL), Dexamethasone Sodium Phosphate Injection, USP (3.2 mg/mL) and 20% contrast in Group 2
  Arms: Group 2 - temsirolimus and dexamethasone injection

SUMMARY:
This is a prospective, multi-center, pilot feasibility study to document the effects of adventitial delivery of temsirolimus or temsirolimus with dexamethasone sodium phosphate injection, USP, after revascularization of femoropopliteal lesions in symptomatic patients with moderate to severe claudication (Rutherford 2-3) or critical limb ischemia (CLI) with rest pain (Rutherford 4). Subjects will be followed for up to 60 months post index procedure.

DETAILED DESCRIPTION:
To begin to assess the safety and effectiveness of Bullfrog Micro-Infusion Device adventitial deposition of temsirolimus or temsirolimus with dexamethasone in maintaining luminal patency and composite safety endpoints in patients with clinical evidence of moderate to severe claudication or critical limb ischemia with rest pain after revascularization of one or more angiographically significant lesion(s) in superficial femoral or popliteal arteries.

ELIGIBILITY:
Inclusion Screening Criteria:

* Age ≥18 years and ≤85 years at study enrollment
* Subject has been informed of the nature of the study, agrees to participate and has signed an IRB-approved consent form
* Subject is ambulatory
* Female subjects of childbearing potential have a negative pregnancy test ≤7 days before the procedure and are willing to use a highly effective method of birth control (See Section 12.2) for one month preceding and 12 months following study treatment
* Subject has documented moderate to severe claudication (Rutherford 2-3) or Critical Limb Ischemia (CLI) with rest pain (Rutherford 4) in the target limb due to arterial stenosis within the superficial femoral and/or popliteal artery
* Life expectancy >2 years in the Investigator's opinion Angiographic Criteria (Target Lesion Definition)
* Target vessel reference diameter ≥3 mm and ≤8 mm
* Single or multiple de novo atherosclerotic or restenotic lesion(s) with ≥70% narrowing in the superficial femoral or popliteal artery meeting the following criteria:

  * The target lesion must be ≤20 cm in total length
  * The target lesion does not have more than 5 cm of contiguous length of intervening normal artery
  * The target lesion does not cross into the common femoral artery or tibeoperoneal trunk
  * The target lesion is located at least 10 mm away from any previously placed stent or graft
* Successful wire crossing (sub-intimal is allowed) and revascularization by balloon angioplasty of the target lesion with less than 30% residual stenosis and run-off in at least one patent vessel into the foot

Exclusion Screening Criteria:

* Subject is already enrolled in another clinical study of systemic drug therapy or another device study that has not completed its primary endpoint
* Subject unwilling or unlikely to comply with visit schedule
* Subjects who are incapable of providing consent and/or incapable of understanding the nature, significance and implications of the clinical trial
* Subject is already receiving, has received in prior 2 months, or is planned in the 6 months after index procedure to receive systemic immunotherapy, chemotherapy, or systemic steroids (however, steroid pre-treatment for contrast allergy, inhaled steroids for asthma treatment or topical steroid uses are allowed)
* Subject is receiving chronic anticoagulation therapy e.g. warfarin (note: chronic antiplatelet therapy, e.g. aspirin and clopidigrel, and procedural anticoagulation therapy, e.g. heparin or bivalirudin, are allowed)
* Subject has a bilirubin level of >1.5xULN
* Recent (<30 days prior to study procedure) myocardial infarction
* Cerebrovascular accident <60 days prior to the study procedure or any history of intracerebral hemorrhage
* Any surgical or endovascular procedure (not including staged revascularization in the target limb, e.g. inflow revascularization prior to index procedure or below-knee revascularization after the index procedure) performed within 14 days prior to the index procedure or planned within 30 days post index procedure
* Planned amputation in the target limb
* Active foot infection or ischemic foot wound
* Inability to receive temsirolimus, dexamethasone or iodinated contrast medium due to labeled contra-indications or known sensitivity reactions
* Estimated glomerular filtration rate (eGFR, calculated from serum creatinine using an isotope dilution mass spectrometry (IDMS)-traceable equation) less than 30 mL/min Angiographic/Procedural Criteria
* Hemodynamically significant inflow lesion (≥50% DS) or occlusion in the ipsilateral iliac artery in which there is failure to successfully treat and obtain a <30% residual stenosis post-revascularization, with bailout stenting as needed (in-flow lesions should be treated prior to treating the target lesion)
* Prior stent placement in target lesion (i.e., in-stent restenosis)
* Target lesion restenosis of any kind within 6 months of a prior intervention
* Use of alternative therapy, e.g. radiation therapy, drug-eluting stents (DES) or drug-eluting balloon/drug-coated balloons (DEB/DCB) as part of the target lesion treatment during the index procedure or during the previous 12 months
* Use of atherectomy devices in the target lesion during the index procedure
* Aneurysm in the target vessel
* Acute thrombus in the target limb
* Heavy eccentric or concentric calcification at target lesion, which in the judgment of the investigator would prevent penetration of the Micro-Infusion Device needle through the vessel wall

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Safety - Freedom from MALE-POD at 30 days | 30 days post intervention
  Freedom from MALE-POD at 30 days
Effectiveness - Primary patency | 12 months post intervention
  Primary patency (adjudicate by angio core lab)
Effectiveness - Freedom from CD-TLR | 12 months post intervention
  Freedom from clinically driven target lesion revascularization (CD-TLR)) at 12 months.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - St. Joseph Hospital of Orange Heart and Vascular Center, Orange, California
  - San Francisco VA Medical Center, San Francisco, California
  - University of Colorado, Denver, Colorado
  - Rocky Mountain Veterans Administration Hospital, Denver, Colorado
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Columbia University Medical Center/NYPH, New York, New York
  - North Carolina Heart and Vascular, Raleigh, North Carolina
  - University Hospital, Cleveland, Ohio
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No